CLINICAL TRIAL: NCT00326339
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Ascending Dose, Dose Ranging Study to Evaluate Up to Three Doses of R935788 in Rheumatoid Arthritis Patients Failing to Respond to Methotrexate
Brief Title: Treatment of Arthritis With Syk Kinase Inhibition (TASKI-1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Elliott Grossbard/SVP Medical Development, Rigel Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-935788-006
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2008-03

CONDITIONS: Rheumatoid Arthritis
Keywords: R935788; Rheumatoid Arthritis; Syk Kinase
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): R788 50 mg PO bid
  Interventions: Drug: R788
- 2 (Experimental): R788 100 mg PO bid
  Interventions: Drug: R788
- 3 (Experimental): R788 150 mg PO bid
  Interventions: Drug: R788
- 4 (Placebo Comparator): Placebo PO bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: R788 — R788 50 mg, 100 mg, or 150 mg PO bid
  Other Names: tamatinib fosdium
  Arms: 1; 2; 3
Drug: Placebo — Placebo PO bid
  Arms: 4

SUMMARY:
This is a Phase II, multicenter, randomized, double-blind, placebo-controlled, ascending dose, dose ranging study to evaluate up to three doses of R935788 (50 mg bid, 100 mg bid and 150 mg bid). Approximately 180 patients who have had rheumatoid arthritis for a minimum of 12 months and who have been receiving a weekly methotrexate (MTX) dose for a minimum of 6 months will be enrolled into the study.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the preliminary efficacy of up to three different dosage regimens of R788 as determined by ACR 20 responder rates at 12 weeks The secondary objectives of this study are to assess the safety of up to three different dosage regimens of R788 as determined by ACR 20 responder rates at 12 weeks, and to assess the general clinical and laboratory safety evaluations throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written informed consent by signing an IRB-approved Informed Consent Form (ICF) prior to admission to this study.
2. Males and females, 18 to 75 years of age, with active RA for at least 12 months (functional class I-III, e.g., not bed or wheelchair-bound) who have been receiving weekly doses of methotrexate (10-25 mg/week) for a minimum of 180 days, and who have been receiving a stable MTX dose of at least 15 mg without any change in route or change in folic acid supplementation for at least 30 days.

   Active RA is defined as the presence of (a)6 swollen joints (28 joint count); AND (b)6 tender joints (28 joint count); AND (c) CRP level > ULN for the central reference laboratory.

   Patient may receive up to 10 mg per day of oral prednisone or steroid equivalent, NSAID therapy, hydroxychloroquine, chloroquine, minocycline, sulfasalazine, and doxycycline. The dose(s) must have been stable for at least 30 days and must not be changed during the washout, screening and treatment periods, unless dictated by tolerability requirements.
3. Females of childbearing potential must be fully informed of the potential for methotrexate and R788 to adversely affect the fetus and must agree to use adequate (2 methods) contraception during the study. These patients must not be lactating and must have a negative urine pregnancy test at the time of randomization and at each laboratory determination.
4. The patient is in otherwise good health as determined by the Investigator on the basis of medical history, physical examination, and laboratory screening tests during the screening period, including the absence of clinically significant findings, such as HIV, HBV or HCV, interstitial pneumonitis or active pulmonary infection, on chest X-ray taken within 6 months prior to screening and a negative TB skin test, or abnormal liver function defined as known ALT >1.2xULN within the past 90 days.
5. In the investigator's opinion, the patient has the ability to understand the nature of the study and any hazards of participation, and to communicate satisfactorily with the investigator and to participate in, and to comply with, the requirements of the entire protocol.

Exclusion Criteria:

1. The patient has a history of, or a concurrent, clinically significant illness, medical condition (other than arthritis) or laboratory abnormality that, in the Investigator's opinion, could affect the conduct of the study (these will be included in an exclusion log).
2. The patient has a history of substance abuse, drug addiction or alcoholism.
3. The patient is unable to abstain from alcohol during the study.
4. The patient has a recent (past 5 years) history of, or treatment for, a malignancy other than basal skin cancer.
5. The patient has received any investigational medication within 30 days prior to admission to the study.
6. Any patient who has received any of the following treatments must abide by the indicated washout period:

   1. oral or injectable gold, azathioprine, penicillamine, anakinra require a 30 day washout period prior to Day 1 dosing
   2. cyclosporine, abatacept, etanercept, infliximab or adalimumab require a 60 day washout period prior to Day 1 dosing
   3. leflunomide requires a 60 day washout period prior to screening, unless the patient has undergone cholestyramine washout at least 30 days prior to Day 1 dosing
   4. cyclophosphamide requires a 180 day washout period prior to Day 1 dosing
   5. Rituxan requires a 180 day washout period and normal CD19 count prior to Day 1 dosing
   6. parenteral or intra-articular corticosteroids require a 30 day washout period prior to Day 1 dosing
7. Patients with the following laboratory abnormalities: ALT > 1.2X ULN, creatinine > ULN, a neutrophil count < 2,500/mm3 or lymphocyte count < 800/mm3, Hgb < 10 g/dL, platelet count < 125,000/mm3 are excluded.
8. Patients should not use CYP3A4 inhibitors from within 3 days of randomization until the end of study. R406 is metabolized by CYP3A4, and ketoconazole increases the R406 AUC of a dose of R788 by approximately 2 fold.
9. Patients should not use CYP3A4 inducers from within 3 days of randomization until the end of the study. Although glucocorticoids are inducers, a stable dose of no more than 10 mg/day is allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2006-08; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The Primary Efficacy parameter is ACR20 response rate at 3 months post dosing. | 12 weeks

SECONDARY OUTCOMES:
ACR 20/50 responses over time | 12 weeks
Disease Activity Score (DAS) at baseline and endpoint | 12 Weeks
Mean changes (SDs) from baseline in Swollen Joint Count (28 joint count) | 12 Weeks
Mean changes (SDs) from baseline in Tender Joint Count (28 joint count) | 12 Weeks
Mean changes (SDs) from baseline in Physician global assessment of disease activity by visual analog scale (VAS) | 12 Weeks
Mean changes (SDs) from baseline in Patient global assessment of disease activity by VAS | 12 Weeks
Mean changes (SDs) from baseline in Patient assessment of pain by VAS | 12 Weeks
Mean changes (SDs) from baseline in HAQ-DI | 12 Weeks
Mean changes (SDs) from baseline in CRP | 12 Weeks
The frequency and severity of Liver Function Test abnormalities, especially ALT and alkaline phosphatase | 12 Weeks
The frequency and severity of hematopoietic cytopenias, principally effects on neutrophil, erythrocyte, and lymphocyte counts | 12 Weeks
The frequency and severity of clinically significant adverse events, especially skin rash, postural dizziness, and alterations in blood pressure and other relevant clinical outcomes | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Grossbard, M.D., Study Director — Rigel Pharmaceuticals; Michael Weinblatt, M.D., Principal Investigator — Brigham and Women's Hospital; Arthur Kavanaugh, M.D., Principal Investigator — University of California, San Diego
Locations (38):
- United States (27):
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - DMI research, Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Arthritis & Osteoporosis Treatment Center, Orange Park, Florida
  - Arthritis Associates Inc., Orlando, Florida
  - Arthritis Research of Florida, Inc., Palm Harbor, Florida
  - Arthritis Research of Florida, Palm Harbor, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - The Center for Arthritis and Rheumatic Diseas, South Miami, Florida
  - Coeur d'Alene Arthritis Clinical Trials, Coeur d'Alene, Idaho
  - The Arthritis Center, Springfield, Illinois
  - MMG Clinical Research, South Bend, Indiana
  - Phase III Clinical Research, Fall River, Massachusetts
  - Michigan Arthritis Research Center, Brighton, Michigan
  - Westroad Medical Group, Omaha, Nebraska
  - NC Arthritis & Allergy Care Center, Raleigh, North Carolina
  - Clinical Research Division, Mayfield Village, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - Altoona Ctr. for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading LLP, West Reading, Pennsylvania
  - Low Country Rheumatology, Charleston, South Carolina
  - Arthritis Clinic, Jackson, Tennessee
  - SCRI, Memphis, Tennessee
  - Austin Rheumatology Research, Austin, Texas
  - Research Across America, El Paso, Texas
  - Center for Arth. & Rheum. Disease, PC, Chesapeake, Virginia
- Mexico (11):
  - Hospital Aranda de la Parra, León, GT
  - Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, JA
  - Hospital Civil de Guadalajara "Dr. Juan I. Menchaca", Guadalajara, JA
  - Clinica para el Diagnostico y Tratamiento de las Enfermedades Reumaticas, S.C., Mexico City, Mexico City
  - Arke Estudios Clinicos, S.A. de C.V., Mexico City, Mexico City
  - Hospital General de Mexico, Mexico City, Mexico City
  - Centro Médico DALINDE, Mexico City, Mexico City
  - Hospital Regional "1° de Octubre", ISSSTE, Mexico City, Mexico City
  - Centro Médico del Instituto de Seguridad Social del Estado de Mexico y Municipios (CMISSEMYM), Metepec, MX
  - Facultad de Medicina y Hospital Universitario "Dr. Jose E. Gonzalez" de la Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León
  - Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, SL